CLINICAL TRIAL: NCT00675246
Title: Antenatal Corticoid Therapy for Fetal Lung Maturation in Late Preterm Pregnancies: a Randomized Controlled Trial
Brief Title: Antenatal Corticoid Therapy for Late Preterm Babies
Acronym: ACTLPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Materno Infantil Prof. Fernando Figueira (Other)
Responsible Party: Ana Maria Feitosa Porto, Instituto Materno Infantil Prof. Fernando Figueira
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CORTICOID001
Record Dates: First submitted 2008-05-07; First posted 2008-05-09 (Estimated); Last update posted 2010-06-09 (Estimated); Status verified 2010-06

CONDITIONS: Hyaline Membrane Disease; Transient Tachypnea
Keywords: corticoid therapy; fetal lung maturation; late preterm; respiratory distress syndrome; neonatal death
MeSH Terms: conditions — Hyaline Membrane Disease; Respiratory Distress Syndrome; Perinatal Death | interventions — Betamethasone; betamethasone acetate phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Antenatal corticoid therapy
  Interventions: Drug: Betamethasone

INTERVENTIONS:
Drug: Betamethasone — IM administration of 12mg of betamethasone each 24 hours (total dose=24mg)
  Other Names: CELESTONE SOLUSPAN (MANTECORP)

SUMMARY:
This study aims to determine the effectiveness of antenatal corticosteroid therapy in late preterm babies. The investigators hypothesis is corticoid accelerates fetal lung maturation even after 34 weeks and reduces risk of respiratory distress syndrome and other neonatal morbidities.

DETAILED DESCRIPTION:
Late preterm babies have important morbidity when compared with term babies, with oxygen requirement and more days of hospitalization. If antenatal corticosteroid therapy is necessary for fetal lung maturation after 34 weeks, it remains to be established. The systematic review with metanalysis in Cochrane Library includes a small number of late preterm babies and no conclusion about effectiveness of corticoid therapy in this setting could be drawn. Our hypothesis is that antenatal corticosteroid therapy is effective to prevent respiratory disease and morbidity in late preterm babies and this study will be carried out to evaluate this question.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy between 34 and 36 weeks
* Confirmed gestational age (LMP, USG)
* Alive fetus
* Imminent risk of preterm delivery

Exclusion Criteria:

* Multiple pregnancy
* Major fetal malformations
* Comproved fetal lung maturity
* Maternal or fetal indication for immediate interruption of pregnancy
* Maternal hemorrhagic syndromes (placenta previa, abruptio placenta)
* Chorioamnionitis
* Chronic use of corticosteroids
* Previous use of corticosteroids for fetal lung maturation in the current pregnancy

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 320 (Estimated)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
neonatal respiratory distress | neonatal period (28 days of life)

SECONDARY OUTCOMES:
during of neonatal hospitalization | neonatal period (28 days of life)
neonatal oxygen requirement | neonatal period (28 days of life)
neonatal sepsis | neonatal period (28 days of life)
neonatal death | neonatal period (28 days of life)

CONTACTS AND LOCATIONS:
Overall Officials: Melania Amorim, MD, PhD, Study Director — Instituto Materno Infantil Prof. Fernando Figueira
Locations (1):
- Instituto Materno Infantil Prof. Fernando Figueira, Recife, Pernambuco, Brazil

REFERENCES:
- [Derived] Porto AM, Coutinho IC, Correia JB, Amorim MM. Effectiveness of antenatal corticosteroids in reducing respiratory disorders in late preterm infants: randomised clinical trial. BMJ. 2011 Apr 12;342:d1696. doi: 10.1136/bmj.d1696. PMID 21487057